CLINICAL TRIAL: NCT04361383
Title: Ultrasound-Guided Erector Spinae Plane Versus Quadratus Lumborum Block For Postoperative Analgesia for Patient Undergoing Open Nephrectomy: A Randomized Controlled Study.
Brief Title: Erector Spinae Plane Versus Quadratus Lumborum Block for Patient Undergoing Open Nephrectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Shereen Elsayed Abd Ellatif, lecturer of anesthesia and surgical intensive care, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 6004-12-4-2020
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-04-21 (Actual); Status verified 2020-04

CONDITIONS: Renal Disease
Keywords: erector spinae plane block; ,Quadratus Lumborum block; open nephrectomy; analgesia
MeSH Terms: conditions — Kidney Diseases; Agnosia | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The patients will be divided randomly by a computer-generated randomization table into three equal groups
Who Masked: Participant, Outcomes Assessor
Masking Description: Double (Participant, Outcomes Assessor)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Placebo Comparator): patients will be operated under general anesthesia.
  Interventions: Other: control group
- QLB group (Active Comparator): patients will receive ultrasound-guided quadratus lumborum block type 3 with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Interventions: Procedure: quadratus lumborum block type 3
- ESPB group (Active Comparator): patients will receive ultrasound-guided erector spinae plane block with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Interventions: Procedure: erector spinae plane block

INTERVENTIONS:
Other: control group — the patient will receive general anesthesia
  Arms: Control group
Procedure: quadratus lumborum block type 3 — patients will receive ultrasound-guided quadratus lumborum block type 3 with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: QLB
  Arms: QLB group
Procedure: erector spinae plane block — patients will receive ultrasound-guided quadratus lumborum block type 3 with 30 ml of bupivacaine 0.25% followed by general anesthesia.
  Other Names: ESPB
  Arms: ESPB group

SUMMARY:
The postoperative pain after open nephrectomy remains a major concern because some patients still demonstrate acute pain that may develop chronic pain that lasts for months following the surgery.

Epidural analgesia is the gold standard for abdominal surgery including for open nephrectomy, however, it has unfavorable side effects such as paresthesia, hypotension, hematomas, an impaired motor of lower limbs and urinary retention that could delay recovery.

Various techniques have tried to replicate the analgesic efficacy of epidural analgesia. They include transversus abdominis plane analgesia (TAP), rectus sheath analgesia (RS), wound infusion analgesia (WI) and transmuscular quadratus lumborum (TQL) analgesia. However, each of these techniques has specific limitations that prevent them from being the analgesic technique of choice for all open abdominal surgeries.

Up to the investigator's knowledge, there is no study done to compare ESPB versus QLB as pre-emptive analgesia in patients undergoing open nephrectomy.

DETAILED DESCRIPTION:
Open surgery remains basic surgery for patients requiring radical or partial nephrectomy and is associated with a high incidence of intense immediate postoperative pain and chronic pain the months following surgery [1]. The physiopathology of acute pain is explained as it is mediated by inflammatory cell infiltration, activation of the pain pathways in the spinal cord, and also reflexive muscle spasm. All of these three mechanisms of acute pain are typically ameliorated during the postoperative recovery [2].

Regional anesthesia techniques are commonly enhanced for pain management in open nephrectomy as they decrease parenteral opioid requirements and improve patient satisfaction [3].

Erector Spinae Plane block (RSPB), first described by Forero et al.,[4] for analgesia in thoracic neuropathic pain, has also been reported for the management of other causes of acute and postoperative pain [5,6,7]. In this ultrasound-guided (USG) technique, a local anesthetic (LA) is applied between the erector spinae muscle and the transverse process of the thoracic vertebra leading to the spread of LA cephalad, caudally and through the paravertebral space [4,5,8].

Quadratus Lumborum block (QLB) was initially described by R.Blanco as an abstract at the annual European Society of Regional Anaesthesia (ESRA) congress in 2007, where the LA was injected at the anterolateral aspect of the QL muscle (type 1 QLB) [9]. Later, J. Børglum used the posterior transmuscular approach by detecting Shamrock sign and injecting the LA at the anterior aspect of the QL (type 3 QLB) [10]. Recently, R. Blanco described another approach by injecting the LA at the posterior aspect of the QL muscle (type 2 QLB), which may be easier and safer as the LA is injected in a more superficial plane, so the risk of intra-abdominal complications and lumbar plexus injuries is less [11]. Finally, the intramuscular QLB (type 4 QLB) was done by injecting LA directly into the QL muscle [12].

The investigators hypothesize that performing ultrasound-guided ESPB block will be more superior to or equal to QLB in providing postoperative analgesia for patients undergoing open nephrectomy under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* BMI ≤ 30 kg/m2
* ASA II and III.
* Elective open nephrectomy under general anesthesia

Exclusion Criteria:

* History of allergy to the LA agents used in this study,
* Skin lesion at the needle insertion site,
* Those with bleeding disorders, sepsis, liver disease, and psychiatric disorders

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2020-04-12 (Actual); Primary Completion 2020-08-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
The 1st time to rescue analgesic | recorded within the first 24 hour postoperatively
  the time to ask for postoperative analgesia is the time from the end of operation to patient reporting VAS ≥ 3.

SECONDARY OUTCOMES:
Visual analogue scale (VAS) | measured at at 1 hour, 2,4,,8,12,18, 24 hour postoperatively
  On a scale of 0-10, the patient will learn to quantify postoperative pain where 0= No pain and 10= Maximum worst pain.
Total dose of rescue analgesia (morphine) | in the first 24 hour postoperatively.
  once the VAS score will be ≥ 3, rescue analgesia in the form of 0.1 mg/kg morphine will be given and the total dose consumed will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of medicine, zagazig university, Zagazig, Elsharqya, Egypt

IPD SHARING:
Plan to Share IPD: Yes
planned after the completion of the study and publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: planned after the completion of the study and publication
Access Criteria: principal investigator

REFERENCES:
- [Background] Gupta V, Yadav SK, Dean E, Vincent P, Walid F, Al Said A. Paediatric laparoscopic orchidopexy as a novel mentorship: Training model. Afr J Paediatr Surg. 2013 Apr-Jun;10(2):117-21. doi: 10.4103/0189-6725.115035. PMID 23860059
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] McCrum CL, Ben-David B, Shin JJ, Wright VJ. Quadratus lumborum block provides improved immediate postoperative analgesia and decreased opioid use compared with a multimodal pain regimen following hip arthroscopy. J Hip Preserv Surg. 2018 Oct 25;5(3):233-239. doi: 10.1093/jhps/hny024. eCollection 2018 Aug. PMID 30393550
- [Background] Niraj G, Tariq Z. Continuous Erector Spinae Plane (ESP) Analgesia In Different Open Abdominal Surgical Procedures: A Case Series. (2018) J Anesth Surg 5(1): 57- 60.
- [Background] Chin KJ, Malhas L, Perlas A. The Erector Spinae Plane Block Provides Visceral Abdominal Analgesia in Bariatric Surgery: A Report of 3 Cases. Reg Anesth Pain Med. 2017 May/Jun;42(3):372-376. doi: 10.1097/AAP.0000000000000581. PMID 28272292